CLINICAL TRIAL: NCT01608594
Title: Neoadjuvant Combination Biotherapy With Ipilimumab (3 mg/kg or 10 mg/kg) and High Dose IFN-Α2B in Patients With Locally/Regionally Advanced/Recurrent Melanoma: a Randomized Safety, Efficacy and Biomarker Study
Brief Title: Neoadjuvant Combination Therapy With Ipilimumab and HighDose IFN-α2b for Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Diwakar Davar (Other)
Responsible Party: Sponsor-Investigator, Diwakar Davar, Assistant Professor of Medicine - Melanoma/Phase 1 Therapeutics, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-063; 11-063 (Other: University of Pittsburgh Cancer Institute)
Record Dates: First submitted 2012-05-26; First posted 2012-05-31 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ipilimumab 10 mg/kg + HDI (Experimental): Ipilimumab 10 mg/kg + standard dose IFN alpha
  Interventions: Drug: administration of ipilimumab10mg/kg
- Ipilimumab 3mg/kg + HDI (Experimental): Ipilimumab 3mg/kg + standard dose IFN alpha
  Interventions: Drug: administration of ipilimumab 3mg/kg + HDI

INTERVENTIONS:
Drug: administration of ipilimumab10mg/kg — Ipilimumab IV infusion:
  * Day 0 (within 1-2 weeks of baseline biopsy) every 3 weeks for 2 doses followed by definitive surgery
  * After surgery recover-y resume at the same dose for 2 additional doses given 3 weeks apart
  * Dose continued 12 weeks later for 4 additional doses given 12 weeks apart
  Interferon Alfa-2b will be given concurrently with ipilimumab. Each patient will receive Interferon Alfa-2b at 20 MU/m²/day intravenously for 5 consecutive days out of 7 every week for 4 weeks, followed by 10 MU/m²/d subcutaneously every other day, 3 times each week for 2 weeks, followed by definitive surgery. After surgery recovery, Interferon Alfa-2b will be resumed at 10 MU/m²/d subcutaneously, every other day three times a week for 46 additional weeks.
  Other Names: MDX-010; MDX-101; BMS-734016; Yervoy
  Arms: Ipilimumab 10 mg/kg + HDI
Drug: administration of ipilimumab 3mg/kg + HDI — Ipilimumab IV infusion:
  * Day 0 (within 1-2 weeks of baseline biopsy) every 3 weeks for 2 doses followed by definitive surgery
  * After surgery recover-y resume at the same dose for 2 additional doses given 3 weeks apart
  * Dose continued 12 weeks later for 4 additional doses given 12 weeks apart
  Interferon Alfa-2b will be given concurrently with ipilimumab. Each patient will receive Interferon Alfa-2b at 20 MU/m²/day intravenously for 5 consecutive days out of 7 every week for 4 weeks, followed by 10 MU/m²/d subcutaneously every other day, 3 times each week for 2 weeks, followed by definitive surgery. After surgery recovery, Interferon Alfa-2b will be resumed at 10 MU/m²/d subcutaneously, every other day three times a week for 46 additional weeks.
  Other Names: MDX-010; MDX-101; BMS-734016; Yervoy
  Arms: Ipilimumab 3mg/kg + HDI

SUMMARY:
The purpose of this study is to evaluate the safety and potential effectiveness of a new treatment for advanced and recurrent melanoma involving the combination of Ipilimumab and IFN-α2b before surgery and to test for biomarker studies in blood and/or tumor to better understand this disease, how best to treat it and what patients should be treated with this combination.

DETAILED DESCRIPTION:
Neoadjuvant therapy allows new insights into melanoma and its biological and immunologic response to therapeutic interventions, such as ipilimumab. Neoadjuvant ipilimumab therapy for high-risk melanoma patients with bulky regional stage IIIB-C lymphadenopathy may result in improved clinical outcome in this group of patients that are more likely to respond to immunotherapeutic interventions and without increased morbidity. Through the design of neoadjuvant trials in which it is possible to obtain biopsy samples, a greater understanding of the dynamic interaction between tumors and the immune system is possible. This should lead to the identification of new targets for the treatment of melanoma and aid in the development of new combinations that may have greater efficacy and acceptable toxicity, to build on the clinical, immunologic, and molecular effect of this therapy for patients with melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, at least 18 years of age
* ECOG performance status 0 or 1
* Histologic diagnosis of melanoma staged:
* Tx or T1-4 and
* N1b, or N2b, or N2c, or N3
* M 0 that may present as any of the following groups:
* Primary melanoma with clinically apparent regional lymph node metastases, biopsy confirmed
* Clinically detected recurrence of melanoma at the proximal regional lymph node(s) basin, biopsy confirmed
* Clinically or histologically detected primary melanoma involving multiple regional nodal groups, biopsy confirmed
* Clinically detected single site of nodal metastatic melanoma arising from an unknown primary, biopsy confirmed
* Patients with intransit or satellite metastases with or without lymph node involvement are allowed if considered surgically resectable at baseline by the treating medical oncologist and surgical oncologist.

NOTE: All patients must be determined to be surgically resectable at baseline to be eligible for this neoadjuvant study.

* Patients must undergo biopsy (punch) or open biopsy (if done as part of a clinically indicated baseline diagnostic procedure) within 14 days of entry into the study. Lymphadenectomy/definitive surgery will be performed after at least 2 and generally not longer than 4 weeks of induction HDI-ipilimumab therapy. Additional delays for definitive lymphadenectomy/surgery are allowed if clinically indicated while awaiting the resolution of potential adverse events from HDI-ipilimumab therapy.
* Patients must have been evaluated by standard-of-care full body imaging studies (CT, PET-CT or MRI) as part of the initial clinical work-up at baseline (no more than 4 weeks prior to study enrollment) and after completion of induction HDI-ipilimumab (at 6-8 weeks after the first dose of ipilimumab/HDI and prior to the definitive lymphadenectomy procedure).
* Required values for initial laboratory tests:
* WBC ≥ 3000/uL
* ANC ≥ 1500/uL
* Platelets ≥ 100 x 103/uL
* Hemoglobin ≥ 10 g/dL
* Creatinine ≤ 1.8 mg/dL
* AST/ALT ≤ 2.5 x ULN
* Bilirubin ≤ 1.5 ULN, (except patients with Gilbert's Syndrome, who must have a total bilirubin less than 3.0 mg/dL)
* No active or chronic infection with HIV, Hepatitis B, or Hepatitis C

Exclusion Criteria:

* Clinical, radiological/laboratory, or pathological evidence of distant metastatic disease.
* Evidence of soft tissue involvement by gross extranodal extension of tumor manifest by fixation to the fascia, or matting of nodal tissue that would compromise surgical resection as determined by the surgical oncologist.
* History of acute diverticulitis, intra-abdominal abscess, GI obstruction and abdominal carcinomatosis which are known risk factors for bowel perforation.
* Any other malignancy from which the patient has been disease-free for less than 5 years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix.
* Autoimmune disease exclusions: a history of inflammatory bowel disease, a history of symptomatic disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [e.g., Wegener's Granulomatosis]); motor neuropathy considered of autoimmune origin (e.g. Guillain-Barre Syndrome).
* Any underlying medical or psychiatric condition, which in the opinion of the Investigator/Sub-Investigator will make the administration of ipilimumab or HDI hazardous or obscure the interpretation of AEs, such as a condition associated with frequent diarrhea.
* Underlying heart conditions if deemed ineligible for surgery by cardiology consult.
* Any non-oncology vaccine therapy used for prevention of infectious diseases (for up to 1 month before or after any dose of ipilimumab).
* Prior treatment with ipilimumab or CD137 agonist or CTLA-4 inhibitor or agonist.
* Prior radiotherapy, chemotherapy, including infusion or perfusion therapy for current disease or any immunotherapy including tumor vaccines, interferon-alfa, interleukins, levamisole or other biologic response modifiers within the past 4 weeks.
* Concomitant therapy with any of the following: IL 2 or other non-study immunotherapy regimens; cytotoxic chemotherapy; immunosuppressive agents; other investigation therapies; or chronic use of systemic corticosteroids; unless discontinued ≥ 4 weeks. A history of occasional use of steroid inhalers is allowed.
* Women of childbearing potential (who:
* Are unwilling or unable to use an acceptable method of contraception to avoid pregnancy for their entire study period and for at least 26 weeks after cessation of study drug, or
* Have a positive pregnancy test at baseline, or
* Are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-05-21 (Actual); Primary Completion 2017-02-14 (Actual); Study Completion 2017-02-27 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 5 years
  To estimate the safety profile of investigational combination biotherapy with standard HDI and ipilimumab at 10 mg/kg and 3 mg/kg

SECONDARY OUTCOMES:
Pathologic response rate | 1 year
  To monitor the pathologic tumor response rate (complete response, microscopic residual disease and macroscopic residual disease) at the time of definitive surgery
Radiologic preoperative response rate | 1 year
  The response rate will be estimated by the percentage of patients who achieve CR, PR or SD by RECIST criteria, with corresponding exact 90% confidence limits being reported for each dose level.
Progression Free Survival | 5 years
  To determine length of time during and after treatment during which the disease does not get worse. Both arms are to be compared.
Overall Survival | 5 years
  the percentage of subjects alive five years after diagnosis or treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Diwakar Davar, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Gorry C, McCullagh L, O'Donnell H, Barrett S, Schmitz S, Barry M, Curtin K, Beausang E, Barry R, Coyne I. Neoadjuvant treatment for stage III and IV cutaneous melanoma. Cochrane Database Syst Rev. 2023 Jan 17;1(1):CD012974. doi: 10.1002/14651858.CD012974.pub2. PMID 36648215
- [Derived] Tarhini A, Lin Y, Lin H, Rahman Z, Vallabhaneni P, Mendiratta P, Pingpank JF, Holtzman MP, Yusko EC, Rytlewski JA, Rao UNM, Ferris RL, Kirkwood JM. Neoadjuvant ipilimumab (3 mg/kg or 10 mg/kg) and high dose IFN-alpha2b in locally/regionally advanced melanoma: safety, efficacy and impact on T-cell repertoire. J Immunother Cancer. 2018 Oct 23;6(1):112. doi: 10.1186/s40425-018-0428-5. PMID 30352626